CLINICAL TRIAL: NCT03821740
Title: Kinesiotaping for Normalizing Scapular Dyskinesis : the Influence on Scapular Kinematics and on the Activity of Scapular Stabilizing Muscles
Brief Title: Kinesiotaping for Normalizing Scapular Dyskinesis
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Camille Tooth, Principal Investigator, University of Liege
Other Study IDs: 1
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Scapular Dyskinesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kinesiotaping — Mc Connel taping and another kinesiotaping technique

SUMMARY:
The 3-dimensional position and orientation of the scapula as well as muscle activation of upper trapezius (UT), lower trapezius (LT) and serratus anterior (SA) of asymptomatic dyskinetic sportspeole will be recorded during shoulder flexion and shoulder abduction, in loaded and unloaded conditions. Participants will be assessed in standard condition and with two differents kinesiotaping techniques.

DETAILED DESCRIPTION:
About 20 dyskinetic asymptomatic people will be involved in the study. The objective will be to compare two different kinesiotaping techniques in normalizing scapular kinematics.

Tridimensional-movement of the scapula and EMG activity of periscapular muscles will be evaluated doing flexion (sagittal plane) and abduction (frontal plane) movements.

EMG acquisitions :

The electromyographic (EMG) signals are collected with Trigno Standard and Trigno Mini wireless sensors (Delsys, Boston, MA, USA) using silver-contact bipolar bar electrodes with ﬁxed 10 mm inter-electrode spacing [49]. Three of the main scapular stabilizing muscles of the shoulder are investigated: upper trapezius, lower trapezius and serratus anterior. Electrodes are placed on the dyskinetic side. In case of bilateral scapular dyskinesis, electrodes are placed on the side where the most important dysfunction was observed. Data are acquired at a sample frequency of 1000 Hz.

Tridimensionnal assessment:

Scapular kinematics is assessed using a three-dimensional motion analysis system, an optoelectronic system based on active markers (Codamotion, Charnwood Dynamic, UK). For that purpose, four Codamotion CX1 units are used, at a sampling of 100 Hz. Fifteen active markers were placed on the skin of the subject on the same side as EMG electrodes: 4 on the thorax, 6 on the scapula, 4 on the arm and 1 on the acromio-clavicular joint.

Procedure :

* Warm up : 2x10 shoulder internal and external rotations
* Maximum voluntary isometric contraction (MVIC)
* 10 mouvements of abduction (frontal plane) + 10 mouvements of flexion (sagittal plane), with and without load in each condition (without kinesiotaping, with a first kinesiotaping technique and with a second kinesiotaping technique). The order of the different conditions will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral scapular dyskinesis (visual evaluation, "yes-no method")
* scapular downward rotation at rest

Exclusion Criteria:

* asymmetry of length of lower limbs
* scoliosis or dorsal hyperkyphosis shoulder surgical history
* shoulder pain, shoulder injury (muscular, osseous, ligamentary, tendinous) or positive tendinous and impingement tests (Jobe, Patte 0°, Patte 90°, Lift off Test, Palm-up Test).

Ages: 18 Years to 35 Years | Sex: Male
Age Groups: Adult
Study Population: Male dyskinetic sportspeople without shoulder pain, from sportsclub in the Province of Liege (Belgium)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
EMG activity of upper trapezius, lower trapezius and serratus anterior | in standard condition and with kinesiotaping (all the same day)
  Measurement with Delsys Trigno (non invasive electrodes)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire d'Analyse du Mouvement Humain, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
Data won't be shared with anyone